CLINICAL TRIAL: NCT00158405
Title: Multicentric Randomised Controlled Trial Assessing the Efficacy of Two Strategies of Structured Treatment Interruption of Highly Active Antiretroviral Therapy (HAART) Compared With a Continuous HAART in HIV- Infected Adults in Abidjan
Brief Title: Randomised Trial of Structured Treatment Interruption of HAART in HIV-Infected Adults in Abidjan (ANRS 1269 TRIVACAN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 1269 TRIVACAN
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-12

CONDITIONS: HIV Infections
Keywords: HIV; Structured treatment interruption; HAART; Sub-saharian africa; Treatment Interruption; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Treatment Interruption; Zidovudine; Lamivudine; efavirenz; Ritonavir; Indinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Structured Treatment Interruption
Drug: Zidovudine (ZDV)
Drug: Lamivudine (3TC)
Drug: Efavirenz (EFV)
Drug: Ritonavir (NRV)
Drug: Indinavir (IDV)

SUMMARY:
Interrupting HAART during limited periods of time ("structured treatment interruption : STI") could entail benefits (better long term tolerance, lower drug-induced viral resistance, lower cost) but also concomitant risks (lower efficacy, higher drug-induced viral resistance). At present, the benefit/risk ratio of STI is unclear. Several STI trials are in progress in industrialised countries. This trial aim at assessing the benefits and risks of two different STI strategies in West Africa.

DETAILED DESCRIPTION:
The objective of this study is to assess the non-inferiority of two strategies of structured treatment interruption (STI) of highly active antiretroviral treatment (HAART) compared with a continuous HAART.

It's a multicentric open labeled randomised non-inferiority trial, which takes place in 5 health care centres in Abidjan, the economic capital city of Cote d'Ivoire

The trial was designed in two phases :

1. Pre-randomisation phase : 840 HAART-naive HIV-infected adults start the following continuous HAART regimen: zidovudine-lamivudine in combination with

   * preferably efavirenz, for HIV-1 infected men, and HIV-1 infected women with an effective contraception and no history of nevirapine-containing p-MTCT (prevention of mother to child transmission);
   * ritonavir-indinavir, for HIV-2 infected patients, women not desiring contraception, and women with a past history of p-MTCT with nevirapine.
2. Trial phase : After at least six months on continuous HAART in the pre-randomisation phase, patients who meet success criteria (CD4 count over 350/mm3, undetectable viral load, absence of current opportunistic infection) are randomised into three arms :

   * Arm 1: Continuous HAART (1 of 6 patients)
   * Arm 2: Fixed STI strategy (3 of 6 patients): immutable periods of 2 months on HAART / 4 months off HAART
   * Arm 3: CD4-guided STI strategy (2 of 6 patients): unlimited interruption of HAART, and then re-introduction/re-interruption guided by the evolution of the CD4 count.

Following the DSMB recommendation, the arm 3 has been discontinued in october 2005. The trial is continuing for patients in the arms 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* 18 years old or more
* CD4 count between 150 and 350 per mm3 (or CD4 percentage between 12.5 and 20 percent)
* no past history of curative antiretroviral therapy
* residence in Abidjan

Exclusion Criteria:

* pregnancy
* severe renal failure
* severe hepatic failure
* severe neuropsychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2002-12; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To assess the non-inferiority at 24 months of two STI strategies of HAART compared with a continuous HAART in terms of :
Percentage of patients with CD4 count over 350 per mm3
Incidence of severe morbidity
Incidence of mortality

SECONDARY OUTCOMES:
To compare at 24 months two STI strategies of HAART with a continuous HAART in terms of :
HIV resistance to antiretroviral drugs
Cost-utility
Compliance to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Anglaret, MD, Study Director — Unité INSERM 593, Université Victor Segalen Bordeaux 2; Christine Danel, MD, Principal Investigator — Programme PACCI, Abidjan; Roger Salamon, Pr, Study Chair — Unité INSERM 593, Université Victor Segalen Bordeaux 2; Emmanuel Bissagnene, Pr, Study Chair — CHU Treichville
Locations (5):
- Côte d’Ivoire (5):
  - Centre de Prise en Charge et de Formation ACONDA, Abidjan
  - Centre de Suivi des donneurs de sang, Centre National de Transfusion Sanguine, Abidjan
  - Centre Intégré de Recherches Biocliniques d'Abidjan, Abidjan
  - Service des Maladies Infectieuses et Tropicales, CHU de Treichville, Abidjan
  - Unité de Soins Ambulatoires et de Conseil, CHU de Treichville, Abidjan

REFERENCES:
- [Background] Moh R, Danel C, Sorho S, Sauvageot D, Anzian A, Minga A, Gomis OB, Konga C, Inwoley A, Gabillard D, Bissagnene E, Salamon R, Anglaret X. Haematological changes in adults receiving a zidovudine-containing HAART regimen in combination with cotrimoxazole in Cote d'Ivoire. Antivir Ther. 2005;10(5):615-24. doi: 10.1177/135965350501000510. PMID 16152755
- [Result] Danel C, Moh R, Minga A, Anzian A, Ba-Gomis O, Kanga C, Nzunetu G, Gabillard D, Rouet F, Sorho S, Chaix ML, Eholie S, Menan H, Sauvageot D, Bissagnene E, Salamon R, Anglaret X; Trivacan ANRS 1269 trial group. CD4-guided structured antiretroviral treatment interruption strategy in HIV-infected adults in west Africa (Trivacan ANRS 1269 trial): a randomised trial. Lancet. 2006 Jun 17;367(9527):1981-9. doi: 10.1016/S0140-6736(06)68887-9. PMID 16782488
- [Result] Danel C, Moh R, Chaix ML, Gabillard D, Gnokoro J, Diby CJ, Toni T, Dohoun L, Rouzioux C, Bissagnene E, Salamon R, Anglaret X; Trivacan ANRS 1269 Trial Group. Two-months-off, four-months-on antiretroviral regimen increases the risk of resistance, compared with continuous therapy: a randomized trial involving West African adults. J Infect Dis. 2009 Jan 1;199(1):66-76. doi: 10.1086/595298. PMID 18986246